CLINICAL TRIAL: NCT06055881
Title: Primary Breast Oligoprogressive Sites Treated With Radiotherapy to Obviate the Need to Change Systemic Therapy (BOSS)
Brief Title: Primary Breast Oligoprogressive Sites Treated With Radiotherapy to Obviate the Need to Change Systemic Therapy
Acronym: BOSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2232; NCI-2023-03208 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-002943 (Other: Mayo Clinic Institutional Review Board); GMROR2232 (Other: Mayo Clinic Radiation Oncology)
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Carcinoma; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Radiosurgery; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic Breast Cancer (Experimental): Breast cancer patients with ER+/PR± (any PR status)/HER2- disease or HER2+ disease (any ER or PR status) will receive radiotherapy that consists primarily of Stereotactic body radiation therapy (SBRT), but at a minimum, it will consist of dose-escalated, moderately hypofractionated radiotherapy (as opposed to conventional fractionation or conventional palliative treatment regimens).
  Interventions: Procedure: Biospecimen Collection; Other: Surveys; Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Blood Sample Collection
Other: Surveys — Patients complete the European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) survey and "Was it Worth It" questionnaire.
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Patients receive stereotactic body radiation therapy (SBRT), metastasis-directed radiation therapy .
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy; stereotactic body radiation therapy
Procedure: Computed Tomography — Undergo CT, MRI and/or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computed Tomography (CT) scan; CT
Procedure: Magnetic Resonance Imaging — Undergo CT, MRI and/or PET/CT
  Other Names: Magnetic Resonance Imaging (MRI); MRI; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MRI Scan; Nuclear Magnetic Resonance Imaging; NMRI; Structural MRI; sMRI
Procedure: Positron Emission Tomography — Undergo CT, MRI and/or PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; Pet Scan; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This study assesses if metastasis-directed radiation therapy (Stereotactic body radiation therapy - SBRT) can delay a change in systemic therapy, and if circulating tumor cells in the bloodstream can help guide treatment options in metastatic breast cancer patients with progressive disease

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histological confirmation of primary breast cancer.
* Patients with metastatic breast cancer and at least 12 months of clinical response to first-line systemic therapy, with the subsequent development of 1-3 extracranial sites of oligoprogressive disease, and who plan for the continuation of the current systemic therapy.

  * NOTE: patients with de novo metastatic disease and those developed metastatic disease after initially localized disease can both be included.

OR

* Patients with metastatic breast cancer and at least 6 months of clinical response to second-line systemic therapy (or further, e.g., third- or fourth-line), with the subsequent development of 1-3 extracranial sites of oligoprogressive disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2.
* Negative urine or serum pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Provide written informed consent.
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
* Willing to provide blood samples for correlative research purposes.
* Receiving radiation therapy as specified in the protocol.

Exclusion Criteria:

* Male patients.
* Nursing or pregnant women.
* Men or women of childbearing potential who are unwilling to employ adequate contraception.
* Patients with triple negative disease (negative for ER, PR, and HER2).
* Active second primary malignancy
* More than 3 extracranial sites of oligoprogressive disease
* Active CNS disease. Patients with asymptomatic and stable, treated CNS lesions (radiation and/or surgery and/or other CNS-directed therapy who have not received corticosteroids for at least 4 weeks) are allowed.

  * Active connective tissue disease that is felt by the treatment team to pose an excess risk of toxicity.
  * Prior radiation that overlaps with the intended treatment volume such that, in the opinion of the patient's Radiation Oncologist, radiotherapy to progressing sites will not be safe.

    * NOTE: patients with some dose overlap with prior radiotherapy that is deemed safe by the patient's Radiation Oncologist can be included in the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2032-05-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from a change in systemic therapy (FCST) - overall | 6 months
  FCST is defined as no change in systemic therapy at 6 months after radiotherapy and patient survival at 6 months after radiotherapy. Treatment failure would indicate that there is no longer stability of systemic therapy (and thereby requires a change in systemic therapy to a different agent).

SECONDARY OUTCOMES:
Freedom from a change in systemic therapy (FCST) - ER+/PR±/HER2- (Subgroup A) | 6 months
  Will assess whether metastasis-directed radiotherapy can result in a clinically significant FCST (defined as for at least 6 months) for patients with estrogen receptor+/progesterone receptor±/human epidermal growth factor receptor 2 negative (ER+/PR±/HER2-) disease. The frequency and percentage for FCST rate will be reported, including the 95% confidence interval.
Freedom from a change in systemic therapy (FCST) - HER2 (Subgroup B) | 6 months
  Will assess whether metastasis-directed radiotherapy can result in a clinically significant FCST (defined as for at least 6 months) for patients with human epidermal growth factor receptor 2 positive (HER2+) disease. The frequency and percentage for FCST rate will be reported, including the 95% confidence interval.
Progression-free survival (PFS) | Up to 5 years
  Will assess the impact of metastasis-directed radiotherapy on PFS in the setting of oligoprogressive breast cancer. PFS is defined as the time from completion of radiotherapy to the first of either disease progression or death from any cause. Medians and 95% confidence intervals will be reported.
Overall survival (OS) | Up to 5 years
  Will explore the impact of metastasis-directed radiotherapy on overall survival (OS) in the setting of oligoprogressive breast cancer. OS is defined as the time from completion of radiotherapy to death from any cause. Medians and 95% confidence intervals will be reported.
Quality of life - EQ-5D-5L | Up to 5 years
  The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a patient-reported outcome measure used to assess health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is rated on a score of 1-5 where 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems/unable to perform the task. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state.
Determine the local control of irradiated, oligoprogressive lesions | Up to 5 years
  This rate will be reported as a percentage with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Roman O. Kowalchuk, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials